CLINICAL TRIAL: NCT01505465
Title: Effects of Perioperative Melatonin on Sleep, Pain, and Confusion After Joint Replacement Surgery
Brief Title: Study of Melatonin on Sleep, Pain, and Confusion After Joint Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2012-032
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Pain; Delirium; Confusion; Sleep
Keywords: Total Knee Replacement; Pain; Confusion; Sleep
MeSH Terms: conditions — Pain, Postoperative; Delirium; Confusion; Pain | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study: Melatonin (Experimental)
  Interventions: Drug: Melatonin
- Control: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 5mg of melatonin will be taken by the subject for 3 nights prior and continuing 3 nights after surgery as tolerated.
  Arms: Study: Melatonin
Drug: Placebo — 5mg of placebo will be taken by the subject 3 nights prior to surgery and continuing 3 nights after surgery
  Arms: Control: Placebo

SUMMARY:
Pain, confusion, and breaks in normal sleep cycles have been challenges commonly faced by patients after undergoing joint surgeries. To address these issues, melatonin, an inexpensive over-the-counter supplement, has shown in previous to help manage sleep disorders, prevent and treat post-operative confusion in patients over 70 years of age, and reduce pain. The purpose of this study is to establish whether melatonin can aid in reducing pain and post-operative confusion and improve sleep quality after total knee replacement

DETAILED DESCRIPTION:
Sleep disruption is a challenge commonly faced by patients and care providers in the perioperative period [1,2] and has been shown to affect postoperative performance after total knee arthroplasty [3] . Postoperative sleep disruption is likely influenced by environmental factors [4] and anesthetic exposure [5,6] and is known to be exacerbated by postoperative pain [7] . In a reciprocal manner, sleep disruption has been shown to exacerbate pain perception [8,9] .

Melatonin is an inexpensive over-the-counter dietary supplement with an established safety profile [10] that has shown promise in managing sleep disorders and amelioration of chronic and acute pain. Evidence suggests that exogenous melatonin can be efficacious in improving sleep disruption in tracheostomized patients in the ICU [11] as well as those experiencing jet lag [12,13] .

Previous studies have found conflicting results regarding the potential for melatonin to improve sleep and pain in the perioperative period [14] . These discrepancies may result from differences in surgical and anesthetic conditions, differences in melatonin dose and administration regimens, variations in study quality, different methods of assessing pain and sleep quality, and different patient populations. There is no consensus as to what dose, duration, and timing of melatonin administration in the perioperative period are most likely to improve sleep quality or quantity. This study was designed to explore the effect of a stable regimen of exogenous perioperative melatonin, administered over 6 consecutive nights, on postoperative pain, sleep quality, and sleep efficiency in patients undergoing total knee arthroplasty under regional anesthesia with sedation. To our knowledge, this study is the first to examine perioperative subjected sleep quality as well as sleep time and efficiency as measured by the validated objective tool of wrist actigraphy in this population.

This study examined the hypotheses that sleep disruption occurs in the context of total knee arthroplasty performed under regional anesthesia with sedation and that perioperative melatonin can modulate pain and sleep disruption after total knee arthroplasty.

1. Gogenur I., Bisgaard T., Burgdorf S., et. al.: Disturbances in the circadian pattern of activity and sleep after laparoscopic versus open abdominal surgery. Surg Endosc 2009; 23: pp. 1026.
2. Kain Z.N., Caldwell-Andrews A.A.: Sleeping characteristics of adults undergoing outpatient elective surgery: a cohort study. J Clin Anesth 2003; 15: pp. 505.
3. Cremeans-Smith J.K., Millington K., Sledjeski E., et. al.: Sleep disruptions mediate the relationship between early postoperative pain and later functioning following total knee replacement surgery. J Behav Med 2006; 29: pp. 215.
4. Lane T., East L.A.: Sleep disruption experienced by surgical patients in an acute hospital. Br J Nurs 2008; 17: pp. 766.
5. Tung A., Mendelson W.B.: Anesthesia and sleep. Sleep Med Rev 2004; 8: pp. 213.
6. Nelson L.E., Guo T.Z., Lu J., et. al.: The sedative component of anesthesia is mediated by GABA(A) receptors in an endogenous sleep pathway. Nat Neurosci 2002; 5: pp. 979.
7. Wylde V., Rooker J., Halliday L., et. al.: Acute postoperative pain at rest after hip and knee arthroplasty: severity, sensory qualities and impact on sleep. Orthop Traumatol Surg Res 2011; 97: pp. 139.
8. Tiede W., Magerl W., Baumgartner U., et. al.: Sleep restriction attenuates amplitudes and attentional modulation of pain-related evoked potentials, but augments pain ratings in healthy volunteers. Pain 2010; 148: pp. 36.
9. Raymond I., Nielsen T.A., Lavigne G., et. al.: Quality of sleep and its daily relationship to pain intensity in hospitalized adult burn patients. Pain 2001; 92: pp. 381.
10. Dietary supplements: a framework for evaluating safety.2005.The National Academies Press Washington, DC
11. Bourne R.S., Mills G.H., Minelli C.: Melatonin therapy to improve nocturnal sleep in critically ill patients: encouraging results from a small randomised controlled trial. Crit Care 2008; 12: pp. R52.
12. Suhner A., Schlagenhauf P., Hofer I., et. al.: Effectiveness and tolerability of melatonin and zolpidem for the alleviation of jet lag. Aviat Space Environ Med 2001; 72: pp. 638.
13. Suhner A., Schlagenhauf P., Johnson R., et. al.: Comparative study to determine the optimal melatonin dosage form for the alleviation of jet lag. Chronobiol Int 1998; 15: pp. 655.
14. Andersen L.P., Rosenberg J., Gogenur I.: Perioperative melatonin: not ready for prime time. Br J Anaesth 2014; 112: pp. 7.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-90 years old undergoing elective, primary total knee replacement
* American Society of Anesthesiologists (ASA) Physical Status I-III
* Epidural anesthesia/Patient Controlled Analgesia candidate

Exclusion Criteria:

* Mental impairment
* Pre-operative use of benzodiazepines, narcotics, or prescription/over-the counter (OTC) sleep aids
* Pre-operative use of calcium channel blockers
* Insomnia
* Recent drug or alcohol abuse
* Psychiatric disorders other than anxiety, including depression
* Diabetes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros G. Memtsoudis, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Ozler M, Simsek K, Ozkan C, Akgul EO, Topal T, Oter S, Korkmaz A. Comparison of the effect of topical and systemic melatonin administration on delayed wound healing in rats that underwent pinealectomy. Scand J Clin Lab Invest. 2010 Oct;70(6):447-52. doi: 10.3109/00365513.2010.506926. PMID 20704520
- [Background] Gitto E, Romeo C, Reiter RJ, Impellizzeri P, Pesce S, Basile M, Antonuccio P, Trimarchi G, Gentile C, Barberi I, Zuccarello B. Melatonin reduces oxidative stress in surgical neonates. J Pediatr Surg. 2004 Feb;39(2):184-9; discussion 184-9. doi: 10.1016/j.jpedsurg.2003.10.003. PMID 14966737
- [Background] Gitto E, Karbownik M, Reiter RJ, Tan DX, Cuzzocrea S, Chiurazzi P, Cordaro S, Corona G, Trimarchi G, Barberi I. Effects of melatonin treatment in septic newborns. Pediatr Res. 2001 Dec;50(6):756-60. doi: 10.1203/00006450-200112000-00021. PMID 11726736
- [Background] Gitto E, Reiter RJ, Cordaro SP, La Rosa M, Chiurazzi P, Trimarchi G, Gitto P, Calabro MP, Barberi I. Oxidative and inflammatory parameters in respiratory distress syndrome of preterm newborns: beneficial effects of melatonin. Am J Perinatol. 2004 May;21(4):209-16. doi: 10.1055/s-2004-828610. PMID 15168319
- [Background] Kucukakin B, Wilhelmsen M, Lykkesfeldt J, Reiter RJ, Rosenberg J, Gogenur I. No effect of melatonin to modify surgical-stress response after major vascular surgery: a randomised placebo-controlled trial. Eur J Vasc Endovasc Surg. 2010 Oct;40(4):461-7. doi: 10.1016/j.ejvs.2010.06.014. Epub 2010 Jul 17. PMID 20638874
- [Background] Kucukakin B, Klein M, Lykkesfeldt J, Reiter RJ, Rosenberg J, Gogenur I. No effect of melatonin on oxidative stress after laparoscopic cholecystectomy: a randomized placebo-controlled trial. Acta Anaesthesiol Scand. 2010 Oct;54(9):1121-7. doi: 10.1111/j.1399-6576.2010.02294.x. PMID 20887414
- [Background] Shigeta H, Yasui A, Nimura Y, Machida N, Kageyama M, Miura M, Menjo M, Ikeda K. Postoperative delirium and melatonin levels in elderly patients. Am J Surg. 2001 Nov;182(5):449-54. doi: 10.1016/s0002-9610(01)00761-9. PMID 11754849
- [Background] Yin YQ, Luo AL, Guo XY, Li LH, Huang YG. Postoperative neuropsychological change and its underlying mechanism in patients undergoing coronary artery bypass grafting. Chin Med J (Engl). 2007 Nov 20;120(22):1951-7. PMID 18067777
- [Background] Karkela J, Vakkuri O, Kaukinen S, Huang WQ, Pasanen M. The influence of anaesthesia and surgery on the circadian rhythm of melatonin. Acta Anaesthesiol Scand. 2002 Jan;46(1):30-6. doi: 10.1034/j.1399-6576.2002.460106.x. PMID 11903069
- [Background] Caumo W, Torres F, Moreira NL Jr, Auzani JA, Monteiro CA, Londero G, Ribeiro DF, Hidalgo MP. The clinical impact of preoperative melatonin on postoperative outcomes in patients undergoing abdominal hysterectomy. Anesth Analg. 2007 Nov;105(5):1263-71, table of contents. doi: 10.1213/01.ane.0000282834.78456.90. PMID 17959953
- [Background] Caumo W, Levandovski R, Hidalgo MP. Preoperative anxiolytic effect of melatonin and clonidine on postoperative pain and morphine consumption in patients undergoing abdominal hysterectomy: a double-blind, randomized, placebo-controlled study. J Pain. 2009 Jan;10(1):100-8. doi: 10.1016/j.jpain.2008.08.007. Epub 2008 Nov 17. PMID 19010741
- [Background] Wilhelmsen M, Amirian I, Reiter RJ, Rosenberg J, Gogenur I. Analgesic effects of melatonin: a review of current evidence from experimental and clinical studies. J Pineal Res. 2011 Oct;51(3):270-7. doi: 10.1111/j.1600-079X.2011.00895.x. Epub 2011 May 26. PMID 21615490
- [Background] Papp M, Litwa E, Gruca P, Mocaer E. Anxiolytic-like activity of agomelatine and melatonin in three animal models of anxiety. Behav Pharmacol. 2006 Feb;17(1):9-18. doi: 10.1097/01.fbp.0000181601.72535.9d. PMID 16377959
- [Background] Yousaf F, Seet E, Venkatraghavan L, Abrishami A, Chung F. Efficacy and safety of melatonin as an anxiolytic and analgesic in the perioperative period: a qualitative systematic review of randomized trials. Anesthesiology. 2010 Oct;113(4):968-76. doi: 10.1097/ALN.0b013e3181e7d626. PMID 20823763
- [Background] Al-Aama T, Brymer C, Gutmanis I, Woolmore-Goodwin SM, Esbaugh J, Dasgupta M. Melatonin decreases delirium in elderly patients: a randomized, placebo-controlled trial. Int J Geriatr Psychiatry. 2011 Jul;26(7):687-94. doi: 10.1002/gps.2582. Epub 2010 Sep 15. PMID 20845391
- [Background] Sultan SS. Assessment of role of perioperative melatonin in prevention and treatment of postoperative delirium after hip arthroplasty under spinal anesthesia in the elderly. Saudi J Anaesth. 2010 Sep;4(3):169-73. doi: 10.4103/1658-354X.71132. PMID 21189854

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Study: Melatonin | Control: Placebo
Started | 25 | 25
Completed | 19 | 18
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study: Melatonin | Control: Placebo | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (65.8) | 61.4 (14.3) | 65.82 (40.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 5 | 12 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Sleep Efficiency
Description: Sleep time change from 96 hours before surgery to 72 hours after surgery
Time Frame: 96 hours before surgery to 72 hours after surgery
Measure: Mean (Inter-Quartile Range); unit: minutes
Arm/Group | Study: Melatonin | Control: Placebo
Number analyzed (Participants) | 19 | 18
minutes | 20 [-25 to 50] | -55 [-100 to -25]

2. Secondary Outcome: Perioperative Effects of Melatonin on Post-operative Pain Scores
Description: A difference in 25% in average pain score at each time point be considered clinically significant.
Time Frame: Up to postoperative day 3
Population: DATA NOT COLLECTED
Arm/Group | Study: Melatonin | Control: Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Melatonin Effects on Delirium During Post-operative Inpatient Stay Based on Clinical Assessment in Patients 65 and Older
Description: A difference of 25% will be considered clinically important.
Time Frame: Up to postoperative day 3
Population: DATA NOT COLLECTED
Arm/Group | Study: Melatonin | Control: Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Melatonin Effects on Daytime Activity
Description: A 20% difference will be considered clinically important.
Time Frame: Up to postoperative day 3
Population: DATA NOT COLLECTED
Arm/Group | Study: Melatonin | Control: Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Melatonin Effects on Patient Controlled Analgesia and Postoperative Narcotic Usage
Description: A 25% in narcotic usage will be considered clinically important
Time Frame: Up to 3 days
Population: DATA NOT COLLECTED
Arm/Group | Study: Melatonin | Control: Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Study: Melatonin | Control: Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes